CLINICAL TRIAL: NCT07098962
Title: Effect of KinesioTaping on Pain at Mediastinal-Thoracic Tube Sites After Cardiac Surgery: A Randomized Prospective Study
Brief Title: KinesioTaping for Thoracic Drain Support
Acronym: KT-Drain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, İsmail DAL, Assistant Professor Literally: Doctor Teaching Member, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KastamonuUnii
Record Dates: First submitted 2025-07-20; First posted 2025-08-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Primary Condition: Pain, Postoperative; Associated Conditions: Cardiac Surgical Procedures, Thoracic Surgery
MeSH Terms: interventions — Athletic Tape; tramadol, dexketoprofen drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping group (Experimental): In this group, KinesioTaping will be applied alongside routine pain management.
  Interventions: Other: Kinesiotaping
- Routine treatment group (Active Comparator): This group will be managed with standard hospital-based painkiller administration.
  Interventions: Drug: Dexketoprofen, tramadol

INTERVENTIONS:
Other: Kinesiotaping — In this group, KinesioTaping will be applied around the thoracic drain sites alongside standard analgesic therapy. This physical therapy technique uses elastic tapes placed on the skin to support healing, reduce pain, and improve patient comfort. The tapes will remain in place for 2-3 days and will be removed together with the drains.
  Other Names: Kinesiotape
  Arms: Kinesiotaping group
Drug: Dexketoprofen, tramadol — Patients in this group will be treated with painkillers consisting of tramadol and dexketoprofen.
  Arms: Routine treatment group

SUMMARY:
This study investigates the effectiveness of KinesioTaping applied around mediastinal and thoracic drain sites in reducing postoperative pain after cardiac surgery. Effective pain management is critical for early mobilization, improved patient satisfaction, and prevention of respiratory complications such as atelectasis. KinesioTaping is theorized to support soft tissue healing, improve circulation, and modulate pain through stimulation of cutaneous mechanoreceptors and fascia adjustment. However, evidence on its efficacy in postoperative settings remains limited. This prospective, randomized controlled trial aims to provide high-quality data on the role of KinesioTaping as a non-pharmacological adjunct for pain management in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Postoperative pain following cardiac surgery is a significant clinical concern that can hinder early mobilization, reduce patient satisfaction, prolong hospital stay, and increase the risk of respiratory complications such as atelectasis and pneumonia. While pharmacological analgesia remains the mainstay of treatment, non-pharmacological adjuncts are increasingly being explored to enhance pain control and reduce reliance on opioids.

KinesioTaping (KT), a method originally developed for musculoskeletal conditions, involves the application of elastic therapeutic tape to the skin with the aim of supporting soft tissue structures, enhancing lymphatic and blood flow, and modulating nociceptive input via stimulation of cutaneous mechanoreceptors. In the context of postoperative care, KT may also help reduce localized edema, support incision sites, and promote a sense of physical stability that contributes to pain relief.

Despite its growing popularity in rehabilitation and sports medicine, the use of KinesioTaping in postoperative settings-particularly in cardiothoracic surgery-remains under-investigated. Limited studies have suggested potential benefits in reducing pain and improving functional outcomes, but current evidence is inconclusive and often methodologically limited.

This prospective, randomized controlled trial aims to evaluate the effectiveness of KinesioTaping when applied around mediastinal and thoracic drain sites in patients undergoing cardiac surgery. The primary objective is to assess postoperative pain levels using validated pain scales (e.g., VAS) in patients receiving KT versus those receiving standard care without taping. Secondary outcomes include opioid consumption, time to ambulation, respiratory function (spirometry or incentive spirometry use), incidence of atelectasis, and patient satisfaction scores.

By providing high-quality evidence on a low-cost, non-invasive, and easily applicable intervention, this study seeks to clarify the potential role of KinesioTaping as an adjunctive tool in postoperative pain management protocols following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery cases
* Patients who are stable until the removal of the chest drain
* Patients who do not experience serious complications such as bleeding or neurological problems

Exclusion Criteria:

* Patients undergoing emergency cardiac surgery,
* Patients with early post-cardiac surgery mortality,
* Patients with conditions requiring reoperation, such as bleeding,
* Patients for whom a pain score cannot be measured, such as neurological complications

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Day 3 Visual Analogue Scale Pain Score | 3 day
  Visual analog scale pain score on the 3th day after cardiac surgery. Pain is defined as no pain (0) or unbearable pain (10).
  0 = No pain, 1-3 = Mild pain, 4-6 = Moderate pain, 7-10 = Severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu Education and Research Hospital, Kastamonu, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
yes
Time Frame: Data will become available persistantly on 2.2.2026.
Access Criteria: Upon reasonable request principal investigator will share the data.